CLINICAL TRIAL: NCT04059588
Title: A Phase I, Dose-escalation Study Investigating the Safety and Tolerability of Intratumoral Injection of an Fc-engineered Anti-CD40 Monoclonal Antibody (2141-V11) in Patients With Cancer
Brief Title: A Study Investigating the Safety and Tolerability of an Immune Treatment in Cancer Patients With Lesions to the Skin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: DKN-0993
Record Dates: First submitted 2019-08-07; First posted 2019-08-16 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Solid Tumor; Cancer of Skin
Keywords: Solid Tumors; Skin lesions; Immunotherapy; CD40 antibody; Cancer; intratumoral; intralesional; metastases; metastasis
MeSH Terms: conditions — Neoplasms; Skin Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Cohorts of 3 to 6 subjects will be sequentially enrolled at progressively higher dose levels of 2141-V 11 using a standard 3+3 dose-escalation design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Injection of 2141-V11 (Experimental): Open label study drug 2141-V11 at escalating doses until MTD is determined, and expansion utilizing the MTD.
  Interventions: Drug: 2141 V-11

INTERVENTIONS:
Drug: 2141 V-11 — intratumoral injection of 2141-V11

SUMMARY:
The purpose of this study is to test the safety and tolerability of 2141-V11 in people who have cancer that does not respond to standard treatment and who have skin lesions (skin tumors) associated with their cancer. The study will also test how the body processes and responds to 2141-V11, and if the study drug has cancer fighting activity in people. The study drug activates a naturally occurring protein called CD40. By activating CD40, cells of the immune system are better able to identify and kill cancer cells.

We are testing if injection of 2141-V11 into metastasis to the skin will be safe and well tolerated, and may result in immune activation in patients with solid tumors that have metastasis to the skin.

DETAILED DESCRIPTION:
This is a Phase 1 open label, dose-escalation study evaluating the safety, pharmacokinetics, pharmacodynamics, immunogenicity, and efficacy of the Fc-engineered variant 2141-V11 in patients with previously treated relapsed or refractory solid tumors and locally advanced or metastatic solid tumors to the skin amenable to intratumoral injection.

There are two parts to the study: a dose-finding stage (Part I), and a dose expansion stage (Part II). Both Part I and Part II of the study will include patients with locally advanced or metastatic cancers of the skin which are not amenable to standard treatment.

A traditional 3 + 3 dose escalation design will be used (Part I). Successive cohorts of participants (3 participants/cohort) will be started on a fixed dose intratumoral injection of 2141V11 at the dose assigned to their cohort. The study drug, 2141-V11, will be dosed once every 3 weeks. The study drug is administered in cycles.

The first group of study participants in Part I will receive the lowest dose of study drug. The next group of study participants will receive the next higher dose. This dosing scheme continues until the maximum tolerated dose is determined. The maximum tolerated dose (MTD) will be defined as 1 dose level below the dose in which DLTs are observed in >33% of the participants.

Participants in Part II of the study will receive the MTD determined from Part 1 (dose escalation) of the study. Part II participants in the study will also receive two vaccinations (KLH and tetanus) to allow monitoring of their immune function.

Participants in both Part I and II can continue to receive cycles of study drug at their assigned dose if they do not experience progression of disease, a serious adverse event, and the study is ongoing.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years old
2. Must have measurable or evaluable metastatic disease (at least more than 1 lesion) as evidenced by physical exam or imaging
3. Must have an identifiable metastatic lesion of the skin, subcutaneous tissue, or lymph node amenable to intratumoral injection. This includes all solid tumors as well as metastatic melanoma and/or melanoma with in-transit metastases.
4. ECOG performance status < 1
5. Histologically confirmed diagnosis of refractory or relapsed metastatic disease
6. Required values for screening laboratory tests:

   * Absolute neutrophil count (ANC) > 1000/mm3 independent of growth factor support
   * Platelets > 75,000/mm3
   * Hemoglobin > 8 g/dl
   * Creatinine clearance > 40 ml/min for the dose-escalation phase, >25 ml/min in dose expansion phase (if safety data from dose escalation indicate this is possible)
   * AST/ALT < 3 x ULN
   * Bilirubin < 1.5 x ULN (except for participants with Gilbert's Syndrome or of non-hepatic origin)
7. Patients must have refractory or relapsed disease and have must have exhausted all standard-of-care therapy for their disease
8. Must be at least 4 weeks since treatment with checkpoint inhibitors or other antibody-based therapy or investigational agents
9. Must be at least 2 weeks since chemotherapy, targeted small molecule therapy, cytokine therapy, or radiation therapy, and be recovered from any clinically significant toxicity experienced during treatment.
10. If sexually active male or female, and participating in sexual activity that could lead to pregnancy, agrees to use two effective methods of contraception (i.e. condom with spermicide, diaphragm with spermicide, hormone-eluting IUD, hormone-based contraceptive with condom). For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug. Men must agree not to donate sperm during and after the study.

    Female study participants of reproductive potential are defined as pre-menopausal women who have not had a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy). Women are considered menopausal if they have not had a menses for at least 12 months and have a FSH of greater than 40 IU/L or if FSH testing is not available, they have had amenorrhea for 24 consecutive months.
11. Women of childbearing potential must have a negative (beta-human chorionic gonadotropin [b-hCG] pregnancy test at screening, as well as a negative pregnancy test prior to each treatment
12. Life expectancy greater than 16 weeks (should be evaluated by a prognostic score, e.g., Royal Marsden score).
13. Able to comply with the treatment schedule as determined by the participant and the LIP

Exclusion Criteria:

1. Concurrent anticancer therapy including investigational agents. This includes topical therapeutic agents.
2. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), risk of pulmonary toxicity, or evidence of active pneumonitis on screening chest CT scan.
3. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
4. Patients with active hepatitis B (defined as having a positive hepatitis B surface antigen (HBsAg) test at screening.
5. Patients with past/resolved hepatitis B virus (HBV) infection (defined as having a negative HBsAg and a positive antibody to hepatitis B core antigen antibody test) are eligible only if polymerase chain reaction is negative for HBV RNA. HBV DNA must be obtained in these patients prior to Cycle 1, Day 1.
6. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
7. Has spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for > 2 weeks prior to screening.
8. Vaccinated with live, attenuated viral vaccines within 4 weeks of enrollment.
9. Known history of human immunodeficiency virus (HIV) or any uncontrolled active systemic infection.
10. Major surgery or a wound that has not fully healed within 4 weeks of enrollment.
11. Treatment with an immunosuppressive regimen of corticosteroids or other immunosuppressive medication (e.g., methotrexate, rapamycin) within 30 days of study treatment. Note: patients with adrenal insufficiency may take up to 5 mg of prednisone or equivalent daily. Topical and inhaled corticosteroids in standard doses are allowed.
12. Severe infections within 4 weeks prior to Cycle 1, Day 1, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
13. Signs and symptoms of infection within 2 weeks prior to Cycle 1, Day 1.
14. Any investigational therapy within 28 days prior to initiation of study treatment. This includes topical or injected agents.
15. Significant cardiovascular disease (i.e., NYHA class 3 congestive heart failure; myocardial infarction within the past 6 months; unstable angina; coronary angioplasty within the past 6 months; uncontrolled atrial or ventricular cardiac arrhythmias.
16. Autoimmune disease including systemic lupus erythematosus, rheumatoid arthritis, multiple sclerosis, Sjogren's syndrome, autoimmune thrombocytopenia, history of uveitis or other autoimmune disease if clinically significant.
17. Patients with clinically active brain metastases are excluded. Patients with stable brain metastasis (with or without intervention) are eligible. Patients with previously irradiated lesions are eligible provided patient is >4 weeks beyond completion of cranial irradiation and >3 weeks of corticosteroid therapy.
18. Known history of leptomenigeal disease, patients with metastases to the brain stem, midbrain, pons, or medulla, and patients with metastases with 10 mm of the optic apparatus (optic nerve and chiasm) will be excluded from the study.
19. Requires anticoagulation with warfarin or equivalent vitamin K antagonists.
20. Has had a pulmonary embolism or any other thromboembolic event within 6 months prior to study entry.
21. Prior toxicities from previous cancer therapy, including checkpoint inhibition, that have not regressed to Grade < 1 severity (NCI CTCAE v4.03, or later versions) within 28 days before Cycle 1, Day 1, with the exception of alopecia.
22. Active hepatitis C are excluded. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
23. Any surgical procedure within less than 14 days of the first receipt of study drug. Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of the need for a major surgical procedure during the study other than for diagnosis.
24. Pregnant or breast feeding
25. Active infection or with a fever >38.5o C within 3 days prior to the first scheduled treatment.
26. Any medical history, including laboratory results, deemed by the investigator to be likely to interfere with their participation in the study, or to interfere with the interpretation of the results, or any social condition that, in the opinion of the Investigator, might pose additional risk to the participant or confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment-emergent adverse events assessed by NCI CTCAE v4.03 | through study completion, an average of 2 years
  Adverse events
Incidence and severity of DLTs reported and their relationship to 2141-V11 administration assessed by NCI CTCAE v4.03 | through study completion, an average of 2 years
  Dose limiting toxities
Change from baseline laboratory assessments and toxicities over time in abnormal Complete Blood Count labs and Complete Metabolic Panel labs assessed by SI laboratory reference ranges | through study completion, an average of 2 years
  Change from baseline laboratory assessments and toxisities over time
Changes from baseline in anti-drug antibody (ADA) responses to 2141-V11 exposure over time | through study completion, an average of 2 years
  Anti-Drug antidoby (ADA) response over time

CONTACTS AND LOCATIONS:
Overall Officials: Juan Osorio, MD, PhD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osorio JC, Knorr DA, Weitzenfeld P, Yao N, Baez M, DiLillo M, Rahman J, Bromberg J, Postow MA, Ariyan C, Robson ME, Ravetch JV. Intratumoral Fc-optimized agonistic CD40 antibody induces tumor rejection and systemic antitumor immunity in patients with metastatic cancer. Res Sq [Preprint]. 2024 Jun 3:rs.3.rs-4244833. doi: 10.21203/rs.3.rs-4244833/v1. PMID 38883779